CLINICAL TRIAL: NCT02123407
Title: Clinical Study on the Harvesting Lymph Nodes With Carbon Nanoparticles for Advanced Gastric Cancer：a Prospective Randomized Study
Brief Title: Clinical Study on the Harvesting Lymph Nodes With Carbon Nanoparticles for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, Peking University, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA2014001
Record Dates: First submitted 2014-04-21; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Advanced Gastric Cancer
Keywords: Advanced Gastric Cancer; Carbon Nanoparticles; Lymph Nodes
MeSH Terms: interventions — Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbon Nanoparticles (Experimental): Carbon Nanoparticles could be used in this arm.The drug is injected into the subserosa of stomach.Injections of 1.0 ml of Carbon Nanoparticles (0.2 ml in each cardinal point adjacent to the lesion) will be performed about 10 minutes before surgery.Then,gastrectomy with D2 dissection will be performed.
  Interventions: Drug: Carbon Nanoparticles
- Gastrectomy with D2 dissection (Active Comparator): Gastrectomy with D2 dissection will be performed in the control arm,no Carbon Nanoparticles or other coloring materials used
  Interventions: Procedure: Gastrectomy with D2 dissection

INTERVENTIONS:
Drug: Carbon Nanoparticles — Carbon Nanoparticles will be injected into the subserosa of stomach around the tumor.Gastrectomy with D2 dissection will be performed after the injection.
  Arms: Carbon Nanoparticles
Procedure: Gastrectomy with D2 dissection — In the control arm,Gastrectomy with D2 dissection will be performed directly,without any coloring materials.
  Arms: Gastrectomy with D2 dissection

SUMMARY:
Carbon Nanoparticles (CNP),with a mean size of 150 nm,can be taken up selectively by lymphatics after injection into the tissue and draining regional lymph nodes are thereby colored black,which may provide surgeons the guidance to lymph node dissection and help them harvest lymph nodes after surgery,especially some small ones. but there was insufficient evidence to justify its efficacy for those purposes.Therefore,the investigators carried out a prospective randomized controlled trial on lymph node vital staining for lymph node dissection and harvesting in advanced gastric cancer to test this idea.

DETAILED DESCRIPTION:
Carbon Nanoparticles (CNP),with a mean size of 150 nm,can be taken up selectively by lymphatics after injection into the tissue and draining regional lymph nodes are thereby colored black,which may provide surgeons the guidance to lymph node dissection and help them harvest lymph nodes after surgery,especially some small ones. but there was insufficient evidence to justify its efficacy for those purposes.Therefore,the investigators carried out a prospective randomized controlled trial on lymph node vital staining for lymph node dissection and harvesting in advanced gastric cancer to test this idea.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and CT confirmed resectable advanced gastric cancer
* No prior treatment
* No metastases

Exclusion Criteria:

* Having allergic reaction
* Pregnant
* R0 resection is not achieved by gastrectomy with D2 lymphadenectomy according to Japanese gastric cancer treatment guidelines 2010 (ver. 3)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
the number of harvested lymph nodes | 1 day after operation

SECONDARY OUTCOMES:
the diameter of harvested lymph nodes | 1 day after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University School of Oncology, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Sasako M, Sano T, Yamamoto S, Kurokawa Y, Nashimoto A, Kurita A, Hiratsuka M, Tsujinaka T, Kinoshita T, Arai K, Yamamura Y, Okajima K; Japan Clinical Oncology Group. D2 lymphadenectomy alone or with para-aortic nodal dissection for gastric cancer. N Engl J Med. 2008 Jul 31;359(5):453-62. doi: 10.1056/NEJMoa0707035. PMID 18669424
- [Background] Catarci M, Guadagni S, Zaraca F, Pistoia MA, Mastracchio A, Trecca A, Ruco L, Carboni M. Prospective randomized evaluation of preoperative endoscopic vital staining using CH-40 for lymph node dissection in gastric cancer. Ann Surg Oncol. 1998 Oct-Nov;5(7):580-4. doi: 10.1007/BF02303825. PMID 9831104
- [Background] Okamoto K, Sawai K, Minato H, Yada H, Shirasu M, Sakakura C, Otsuji E, Kitamura K, Taniguchi H, Hagiwara A, Yamaguchi T, Takahashi T. Number and anatomical extent of lymph node metastases in gastric cancer: analysis using intra-lymph node injection of activated carbon particles (CH40). Jpn J Clin Oncol. 1999 Feb;29(2):74-7. doi: 10.1093/jjco/29.2.74. PMID 10089947
- [Background] Siewert JR, Kestlmeier R, Busch R, Bottcher K, Roder JD, Muller J, Fellbaum C, Hofler H. Benefits of D2 lymph node dissection for patients with gastric cancer and pN0 and pN1 lymph node metastases. Br J Surg. 1996 Aug;83(8):1144-7. doi: 10.1002/bjs.1800830836. PMID 8869330